CLINICAL TRIAL: NCT00469196
Title: Tomotherapy Treatment for Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU-11-0077 / 22933
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Mesothelioma
Keywords: mesothelioma; tomotherapy
MeSH Terms: conditions — Mesothelioma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Tomotherapy — 40 Gy in 15 fractions, at one fraction per day. Dose will be prescribed to the 95% isodose line.

SUMMARY:
Mesothelioma is an incurable cancer involving the lining of the lung. Patients usually suffer progressive symptoms of shortness of breath and chest pain, until they ultimately succumb to the disease. While a very small number of patients qualify for aggressive treatment with surgery, chemotherapy and radiation, and enjoy long-term survival, the vast majority of patients have incurable disease. The treatment options currently available, including chemotherapy and radiation treatment, are only modestly effective at alleviating symptoms and improving life expectancy. This trial explores the use of new radiation technology (tomotherapy), to treat mesothelioma more aggressively than has been possible before. Tomotherapy's ability to treat unusual shaped tumours, particularly when they are wrapped around sensitive normal tissues (the lung), enable higher doses of radiation to be used and this may improve its effectiveness. We will treat 17 patients with tomotherapy and assess the breathing, symptoms, and quality of life of the patients before and after treatment

DETAILED DESCRIPTION:
Background

Malignant mesothelioma of the pleura is one of the most challenging diseases to treat in oncology. It is often associated with previous exposure to asbestos many years in the past with the mean latency period between asbestos exposure and the development of mesothelioma being approximately 48 years. The disease most commonly presents in the fifth to seventh decade of life, and the natural history is one of relentless progression and eventual death in nearly all patients. It can metastasize to regional nodes and/or distant sites, but most of the morbidity and mortality comes from local disease in the chest, causing progressive constriction, and death from pulmonary insufficiency or infection. Common clinical manifestations can include pleural effusions, superior vena cava obstruction, dysphagia, and laryngeal nerve palsy. Median survival rates are generally less than one year from the time of diagnosis, although there may be a small subset of patients with more indolent disease that have longer survival durations. Patients generally suffer from significant symptoms over the course of their illness, particularly progressive dyspnea and chest pain.

Treatment options with mesothelioma

The treatment of mesothelioma has been characterized by disappointment. The only form of "curative" treatment that has been attempted is a combination of surgery (extrapleural pneumonectomy), chemotherapy, and radiation treatment to the hemithorax. This was described by Sugerbaker, who reported 5-year survival rates of 22% of 120 patients treated. Unfortunately, this approach is only possible for early stage disease (clinical stage I with no nodal involvement) in the absence of comorbid medical illness, and the vast majority of patients present with disease too advanced to consider this approach.

Role of radiotherapy in malignant mesothelioma:

Radiation therapy has been used with both radical and palliative intent. Radical treatment with tumoricidal doses is difficult to achieve with conventional treatment machines due to the dose limitations of normal tissues. The liver, heart, stomach, and normal lung tissue is routinely encompassed within the planning target volumes and all of these tissues have tolerances below the doses necessary to control disease. Curative (adjuvant) treatment has also been given after extrapleural pneumonectomy, which does not have the problem of underlying lung to deal with, but the other nearby normal structures are still difficult to avoid.

A main component of the problem in both curative and adjuvant radiotherapy is the presence of chest wall and diaphragm motion during radiotherapy. Breathing motion affects the chest wall and diaphragm primarily, two of the principal targets in mesothelioma. Maneuvers such as breath holding and respiratory gating, which have shown limited success in lung cancer radiotherapy, are more difficult in mesothelioma due to the presence of significant dyspnea and pain in a majority of patients. Clearly any attempt to treat the thoracic pleura with high-dose radiotherapy must either limit or at least account for this organ motion.

The published results from treating mesothelioma with primary radiotherapy have been suboptimal. High dose treatment to the hemithorax using conventional linear accelerators has typically resulted in complete loss of function of the underlying lung, with no survival benefit over palliative radiotherapy or no treatment. However, studies have suggested that specific symptoms can be effectively palliated with focused radiation treatment. Gordon et al reviewed 29 courses of palliative radiotherapy in 19 patients, with varying dose/fractionation schedules. Overall 11/29 treatment courses resulted in complete, "substantial", or partial relief of symptoms. Furthermore, palliation of symptoms strongly correlated with doses over 40 Gy, suggesting a dose-response relationship. Other investigators have shown effective palliation with lower doses. Davis et al treated patients with 20-30 Gy in 4-10 fractions, with response rates of 60-68%. De Graaf-Strukowska showed 50% pain response rates in patients treated to a mean dose of 36 Gy at a minimum of 4 Gy per fraction.

These studies suggest that although radiation is an effective treatment modality against mesothelioma, the technical difficulties in treating the pleural space effectively limit the risk-benefit ratio.

Helical tomotherapy as a technique to treat mesothelioma

Tomotherapy is a relatively new technology which delivers intensity modulated radiation in a helical fashion, much like a spiral CT scan. Because treatment is given from all angles around a patient, the resulting dose distributions are highly conformal and effectively reduce nearby normal tissues. Mesothelioma was identified early in tomotherapy's development as an ideal site for this technology, since the target volume is extremely difficult to treat using conventional techniques but well suited to the tangential beams of tomotherapy. A test plan using tomotherapy to "treat" a sample patient resulted in excellent dose coverage of the pleural disease with acceptable dose delivered to the ipsilateral and contralateral lungs [unpublished data]. Nevertheless, these test plans were designed on static systems in the absence of respiratory motion, so the feasibility of treatment on breathing patients remains unproven. Tomotherapy is currently in routine clinical and research use in several centres across North America, including the Cross Cancer Institute where it was commissioned in 2003.

Study Objectives

Primary Endpoint

The primary endpoint is disease-specific symptom control rate post-treatment, based on Palliation Index [Gordon 1982].

Secondary Endpoints

Overall survival Radiographic response rate at 3 months post-treatment Quality of life scores (QLQ-L30) at 1-, 3- and 6-months post-treatment Acute and subacute toxicity of treatment Feasibility of using cine-MR, using 3T-MRI, to define target volumes in mesothelioma Performance status at 1-, 3- and 6-months post-treatment Pulmonary function test results at 1-, 3- and 6-months post-treatment

Study Design

Description of the study

This is a single institution single-arm phase II study, assessing the efficacy of tomotherapy-delivered radiation in patients with symptomatic mesothelioma. Patients are treated with radiation alone (no concurrent chemotherapy), and assessed for symptoms and performance status post-therapy.

Duration of study

Based on our statistical analysis (see below), we will require 14 analyzable patients. With a potential drop-out rate of 20%, we will accrue 17 patients in total. Assuming a possible accrual rate of one patient every 1-2 months, it may take 24-34 months to complete the accrual process.

Selection of Patients

Eligibility Criteria

Histologic diagnosis of pleural mesothelioma Age>18 Life expectancy > 4 months Able to breathe comfortably in a supine position for periods of approximately 20 minutes (with or without supplemental O2) Has denied treatment with pemetrexed chemotherapy, or has evidence of progressive or refractory disease on treatment with pemetrexed.

Not eligible or has declined aggressive multimodality (surgical) management for early-stage disease Signed informed consent CT scan of chest performed within 6 weeks of study entry

Ineligibility Criteria

Any contraindications to thoracic radiotherapy In the judgment of the treating physician, inadequate pulmonary reserve to tolerate the proposed radiotherapy.

Unable to perform shallow breathing in a manner to make tomotherapy delivery possible Presence of symptomatic distant metastatic disease

Pre-treatment imaging

Pre-simulation imaging is required as part of this study in order to quantify the extent of chest wall and diaphragm movement during the breathing cycle. Two approaches to this analysis are acceptable: MR imaging (using the 3T MRI in the CBIAR facility) or CT/fluoroscopy (using equipment in the radiation oncology department). The decision on which technique to use will depend on the status of the MRI equipment for breathing assessment at the time of patient accrual.

Patient follow-up and evaluations

Baseline 1- month 3-months 6-months History/physical a a a a PFTs a a a a PS a a a a Palliation index a a a a QOL a a a a CT chest a a Planning MR imaging a

Statistical considerations

The number of patients required is based on the estimated efficacy of the proposed treatment regimen and the desired level of statistical significance. The table below indicates the relationship between these factors and the number of patients required:

Response rate Required "n" P-value 0.05 59 0.048 0.10 29 0.047 0.15 19 0.046 0.20 14 0.044 0.25 11 0.042 0.30 9 0.040

Based on the estimated response rate of the proposed treatment (ability to achieve some relief of symptoms), if "n" patients are treated then at least one patient will demonstrate a measurable response more than 95% of the time. In this study, an efficacy of 20% was chosen as a worst-case scenario, below which the treatment would likely not be offered for palliation. Therefore, 14 evaluable patients will be required to refute the null hypotheses of the treatment being ineffective.

If the true efficacy rate is higher, then the likelihood of a false negative result is lower, and an estimate of the true response rate can be learned.

ELIGIBILITY:
Inclusion Criteria:

* histologic mesothelioma
* refused/ineligible for surgery or chemotherapy
* life expectancy >3 months

Exclusion Criteria:

* contraindications to thoracic radiotherapy
* unable to lie flat for duration of radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 6 months
  Disease-specific symptom control rate post-treatment, based on Palliation Index [7].

SECONDARY OUTCOMES:
Breathing Function | 6 months
  Pulmonary function test results at 1, 3 and 6 months post treatment
Survival/Response Rate | 6 months
  performance status at 1, 3 and 6 months post treatment; and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Rufus Scrimger, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada